CLINICAL TRIAL: NCT04275258
Title: Collaborative Opioid Taper After Trauma: Preventing Opioid Misuse and Opioid Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Harborview Injury Prevention and Research Center (Other)
Responsible Party: Principal Investigator, Mark Sullivan, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00008440; 1 R49CE003087-01-00 (Other Grant/Funding Number: CDC); 1R49CE003087-01 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Opioid Use; Pain, Postoperative; Opioid Use, Unspecified; Trauma; Opioid-use Disorder
MeSH Terms: conditions — Pain, Postoperative; Wounds and Injuries; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will use a randomized controlled trial design. Patients taking opioids prior to trauma are at an increased risk for adverse opioid outcomes, therefore we will stratify randomization so that the intervention and control groups are half opioid exposed and half opioid naïve at the time of trauma, Patients with any prescription opioid use in the 30 days prior to trauma will be considered opioid-exposed, while those with no prescription opioid use in the prior 30 days will be considered opioid naïve.
Who Masked: Outcomes Assessor
Masking Description: The team member that coordinates subject's follow-up survey completion after hospital discharge will be masked.
  Team members involved with outcome analysis will be masked.
  .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Subjects will receive standard trauma discharge plan and no more than a 2-week supply of opioids. Subjects will complete surveys at baseline, 12-week, and 24-week post hospital discharge. In addition, subjects will receive:
  * A face-to-face meeting prior to discharge where the PA will discuss with the subject their individualized pain management plan and individualized opioid taper plan.
  * PA will contact subject on the phone within the first week after hospital discharge to ensure subject plans to follow up with PCP and to troubleshoot any subject concerns related to pain management.
  Interventions: Other: Provide assistance to subject's rural PCP pertaining to subject/patient pain management goals and opioid taper plan
- Control group (No Intervention): Subjects will receive standard trauma discharge plan and no more than a 2-week supply of opioids. Subjects will complete surveys at baseline, 12-week, and 24-week post hospital discharge.

INTERVENTIONS:
Other: Provide assistance to subject's rural PCP pertaining to subject/patient pain management goals and opioid taper plan — PA checks in with PCP at 1,2,4,8, 12, 16, and 20 weeks post hospital discharge by secure e-mail, fax or phone to provide opioid taper and pain management guidance until patient has tapered off opioids or returned to pre-trauma doses. PCP may contact PA whenever needed.
  If PCP requests assistance or reports deviation from the planned opioid taper, PA will provide individualized consultations, which may include a revised taper plan and/or adjunctive therapy recommendations.
  If there is continued deviation from the planned taper, the PA will facilitate a UW TelePain multidisciplinary telemedicine consultation.
  The collaborative pain care and opioid taper intervention ends at 20 weeks.
  Arms: Intervention group

SUMMARY:
The investigators will enroll 100 participants using a randomized control trial design to implement and evaluate an individualized opioid taper program supporting rural Primary Care Physicians (PCPs) caring for patients with moderate to severe trauma discharged on opioids. This study will link a trauma center Physician Assistant (PA) with rural PCPs to facilitate pain care and the individualized opioid taper. The investigators seek to improve patient's pain and opioid outcomes and support the PCPs who assume care for these complex patients after hospital discharge.

Our long term goal is to provide a service that will help trauma patients as they go back into primary care and into pain- and opioid-free living.

DETAILED DESCRIPTION:
This study explores the feasibility, efficacy, and potential sustainability of a collaborative pain care/opioid taper strategy for patients discharged to a rural PCP practice on opioids after hospitalization for moderate to severe traumatic injury.

The randomized control study design will provide important pilot data on the efficacy of opioid taper in the context of engaged pain management care at the PCP level when the PCP is supported by expert consultation and has broad implications for patient and clinician education.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years old
2. Injury Severity Score of 9 or greater
3. Resident of Washington state
4. Will be discharged to a rural zip code outside of king county.
5. Glasgow Coma Score of 15
6. Able to read, speak, and write English or Spanish.
7. Has an identifiable PCP or willing to accept referral to a local Federally Qualified Health Center (FQHC)
8. Has an insurer included in the All Payer Claims Database
9. Planned to be discharged on opioid medication
10. Planned to be discharged back to the community

Exclusion Criteria:

1. Less than 18 years old
2. Injury Severity Score less than 9
3. Patient is in judicial custody
4. Resident of a state other than Washington
5. Will not be discharged to a rural zip code outside of king county.
6. Evidence of OUD diagnosis (including using heroin or other illicit opioids in the past month, a DSM-5 OUD diagnosis, or evidence of taking methadone, buprenorphine, or naltrexone).
7. Currently in cancer treatment or enrolled in palliative or hospice care
8. Residing in a nursing home or assisted living facility
9. Using any implanted device for pain control
10. Self-report of heroin or other illicit opioid use in the past month
11. Psychotic symptoms, psychiatric hospitalization or suicide attempts in the past year (including current admission).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary pain outcome: Pain, Enjoyment, General Activity (PEG) | 24 weeks
  Patient reported 0-10 pain severity, enjoyment of life interference, general activity interference total score
Primary opioid outcome: percent of patients at or below their pre-trauma opioid daily dose | 24 weeks
  Percent of patients at or below pre-trauma opioid dose

SECONDARY OUTCOMES:
PROMIS-29 health status | 24 weeks
  Self-reported health status: physical function, anxiety, depression, fatigue, sleep, social. role satisfaction, pain interference, pain intensity Score range 29-150. HIgher scores better on positively worded items: physical function, social role satisfaction. Higher scores worse on negatively worded items: anxiety, depression, fatigue, sleep, pain interference, pain intensity
Illicit drug use | 24 weeks
  DAST-10 Drug screening questionnaire. Ten yes/no items scored 0 or 1. Score range 0-10
Problem alcohol use | 24 weeks
  AUDIT-C Alcohol Use Disorders Indentification Test
Past-month cannabis use | 24 weeks
  Monitoring the Future cannabis frequency questions
satisfaction with pain care | 24 weeks
  HUNT3 study- patient experience with PCP. 3 items scored 0-10. Range 0-30

OTHER OUTCOMES:
Feasibility | 24 weeks
  Percent of eligible patients approached, consented, assessed and contacted after discharge. Percent of primary care providers reached for at least one contact
Sustainability | 24 weeks
  Cost comparison of implementing collaborative opioid taper support vs. control
Fidelity | 24 weeks
  Degree to which the interventionist PA delivered the program as intended
Adoption | 24 weeks
  Uptake of the collaborative care intervention by PCPS (% of PCPs making contact)
Acceptability of Intervention Measure (AIM) | 24 weeks
  Level of satisfaction with the collaborative opioid taper program- 4 item measure range 4-20
Intervention Appropriateness Measure (IAM) | 24 weeks
  Perceived fit of the collaborative taper program with primary care practice4 item measure range 4-20
PCP Feasibility of Intervention Measure (FIM) 4 item measure range 4-20 | 24 weeks
  PCP ease of engagement during collaborative care contacts

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sullivan, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sullivan MD, Katers L, Wang J, Arbabi S, Tauben D, Baldwin LM. A randomized trial of collaborative support for opioid taper after trauma hospitalization. Subst Abuse Treat Prev Policy. 2024 Jun 24;19(1):33. doi: 10.1186/s13011-024-00613-x. PMID 38915106